CLINICAL TRIAL: NCT04374227
Title: The Effect of Osteopathic Manipulative Treatment (OMT) on Proprioception in Adults: A Pilot Study
Brief Title: The Effect of Osteopathic Manipulative Treatment (OMT) on Proprioception in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Des Moines University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2019-26
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Osteopathy in Diseases Classified Elsewhere
MeSH Terms: interventions — Manipulation, Osteopathic

STUDY DESIGN:
Intervention Model Description: The subjects were randomized into treatment or control groups. The treatment group for week 1 completed two measurements (before and after) and one treatment. Week 2 the treatment group received a treatment. Week 3 the treatment group received a treatment. Week 2 they completed one measurement. The control group completed two measurements and an assessment during week 1. They completed an assessment during weeks 2 and 3, and then completed a measurement during week 4.
Who Masked: Outcomes Assessor
Masking Description: The person running the force plate and its analysis was blind to who was in the treatment group and who was not because the analysis and treatments were given in different rooms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): The treatment group received three osteopathic manipulative treatments once a week for three weeks. The osteopathic manipulative treatment was a full body treatment based upon Dr. Zink's model of a common compensatory pattern.
  Interventions: Procedure: Osteopathic Manipulative Treatment
- Control Group (No Intervention): This group received an osteopathic structural exam once a week for three weeks without any treatment performed.

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment — Body regions that were treated included head, cervical, thoracic, ribs, lumbar, pelvis, sacrum, lower extremity, and upper extremity.
  Arms: Treatment Group

SUMMARY:
Participants will be recruited from the Des Moines University community and randomized into treatment and control groups. The treatment group will undergo three treatments one week apart. The control group will have an osteopathic structural exam without treatment. During the first treatment weeks both groups will undergo balance testing on a force plate pre and post intervention. Additional balance testing will take place one week after last intervention. Six variables will be compared between groups used a linear mixed model analysis.

DETAILED DESCRIPTION:
Participants will go through an informed consent process, fill out a screening questionnaire and will undergo neurological testing. If there are any abnormalities in their neurological testing or they meet exclusion criteria, they will not be included in the study. The neurological testing will include reflex testing, sensation testing, strength testing, and coordination and balance tests.

Participants will then be randomized into 2 groups. One control and one treatment.

Each group will have their balance measured using the portable force plate. Participants will be tested on both feet with arms crossed and eyes open for 60 seconds, and both feet with arms crossed and eyes closed for 60 seconds. Then they will be given 15 seconds to practice standing on the force plate on only their right leg with eyes open and arms crossed. The investigators will then test their balance on their right leg with arms crossed and eyes open for 30 seconds. They will be given 15 seconds to practice standing on their right leg with their arms crossed and eyes closed, and then will have their balance tested on their right leg with arms crossed and eyes closed for 30 seconds. The same sequence of events will take place for the left leg as their right leg. This sequence of measurements will take place at the beginning and end of their first treatment visit. For the standing test with eyes closed and all single leg tests someone will be standing beside the force plate with an arm and either side of the participant to prevent the participant from falling and hurting themselves.

The force plate calculates the center of mass of the participant, the area that is covered by the center of mass, the length of the path of center of mass, the velocity of its motion, and the maximum sway in the x and y planes.

During the single leg tests, the investigators will also record the time of when the participant brings the other foot down, touches the two legs together, or if the sternum becomes outside the borders of the pelvis, if they do lose their balance The test duration will be 30 seconds, as stated previously.

Between the two balance tests, the treatment group will receive a full-body osteopathic manipulative treatment according to the Common Compensatory Pattern (CCP). CCP is a treatment approach developed by Dr. Zinc that addresses the transition areas of the body. The treatment will be given by one of the four fellows under supervision by a licensed physician and last 10-20 minutes. The treatment will include the following body regions:

Occipito-atlantal Joint Thoracic Inlet Thoraco-lumbar shift Lumbo-pelvic roll Ribs Sacrum Pelvis Upslip Upper extremity Lower extremity

The fellows will diagnose somatic dysfunctions within these body regions, treat, and reassess to make sure the somatic dysfunctions are resolved. The physician will perform a spinal sweep and side-to-side height assessments before and after treatment to verify there was improvement in somatic dysfunctions.

After the treatment, the treatment group will walk around the perimeter of the lab for 5 minutes before retesting their balance.

The control group will be asked to lay on an OMM (Osteopathic Manual Medicine) treatment for 15 minutes. They will then walk around the perimeter of the lab for 5 minutes before retesting their balance.

The treatment group will come for five visits. The first visit will include the informed consent and neurological exam. The second visit will include a balance measurement, a treatment, and a follow-up balance measurement immediately after the treatment. The next two visits will consist only of osteopathic treatments. Each visit will be spaced one week apart. The participant will come back a week after their last treatment and complete follow-up balance testing.

The control group will have a total of five visits. They will have the same initial visit as the treatment group with informed consent and neurological exam. Their second visit will consist of a balance measurement, have somatic dysfunctions be diagnosed, yet not be treated and have an immediate follow-up measurement. The third and fourth visits will consist of diagnosing somatic dysfunctions without any treatment. The last visit will consist of a follow-up balance testing. Each of these visits will be one week apart.

The data from the force that will be used includes area that the center of mass covers, length of pathway of center of mass, velocity of the center of mass, medial-lateral sway, and anterior-posterior sway. The investigators will also use the length of time participants were able to stand on one leg without losing their balance (without moving their knee or chest outside of their midline, their foot leaving the platform, touching their opposite foot to the ground, or letting their legs touch).

Summary descriptive statistics will be first obtained for the selected variables and demographics covariates as appropriate. For a particular variable, the change between pre- (or baseline) and post- treatment during the first week reflects the immediate treatment effect while the difference between the pre-treatment baseline and the last measurement during week 4 represents the long-term lasting accumulative effect. The data bear the characteristics of repeated measurements on the same study participants since more than one measurements are taken on the same study participant over time. Thus, it is usually plausible to assume the measurements on the same individual subjects are correlated. Ignoring the covariance between such measurements may result in erroneous statistical inference, and avoiding it by data transformation may result in inefficient statistical inference. The statistical technique of linear mixed model allows the covariance structure to be integrated into the modeling while accounting for the randomness of the study subjects. Thus, the data will be analyzed separately for each variable with a linear mixed-effect model with repeated measures design to assess the OMT effects on the balance measurement metrics over time. In the model fitting process, several candidate covariance structures will be selected and evaluated according to the experimental design (i.e., unequal spacing of the time points but with the same time points across the study participants, within-subject correlation over time and convergence of model fitting), out of which one optimal covariance structure will be selected by the Akaike information criterion (AIC) criteria. On the basis of the chosen models for the respective variables, statistical contrasts will be set up to compare the mean values of variable measurements between time points to assess the immediate and long-term effects of OMT treatment. Tukey procedure for the multiple testing adjustment will be used to compute the adjusted p-value in case of need.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18-40 years old
* Have the ability to give consent
* Be able to bare weight on both feet

Exclusion Criteria:

* had manipulation performed by a D.O., physical therapist, or chiropractor in the last two months,
* had surgery in the six months
* had broken or fractured a bone in the last six months
* have an abnormal neurological exam
* cerebellar dysfunction or ataxia
* has a condition that impairs balance (including orthostatic hypertension,otoneurologic conditions, or arrhythmias)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-10-16 (Actual); Primary Completion 2019-11-21 (Actual); Study Completion 2019-11-21 (Actual)

PRIMARY OUTCOMES:
Length of pathway of center of mass | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  the center of mass of the participant is tracked on the force plate and the overall length it travels will be recorded
area covered by center of mass | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  the center of mass of the participant is tracked on the force plate and its total area covered was measured
velocity of center of mass | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  the center of mass of the participant is tracked on the force plate and the velocity at which that point moved was measured
medial-lateral sway | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  the center of mass of the participant is tracked on the force plate and the amount of lateral movement the point had was measured
anterior-posterior sway | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  the center of mass of the participant is tracked on the force plate and the amount of front-to-back movement the point had was measured
Time | 60 seconds for two leg testing, 30 seconds for single leg testing, timing may de different if participant fell
  we measured the amount of time participants were able to stand upright without touching the ground or having one leg touch the other in the single-leg tests

CONTACTS AND LOCATIONS:
Locations (1):
- Des Moines University, Des Moines, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-01): https://cdn.clinicaltrials.gov/large-docs/27/NCT04374227/Prot_SAP_000.pdf